CLINICAL TRIAL: NCT00391365
Title: Treatment Outcomes for Ankle Arthritis
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Orthopaedic Associates of Michigan (Grand Rapids, MI) (Unknown); Orthopedic + Fracture Specialists, Portland, OR (Other); Minnesota Orthopedic Sports Medicine Institute Twin Cities Orthopedics (Edina, MN) (Unknown)
Responsible Party: Sponsor
Other Study IDs: F4513-R
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis
Keywords: ankle osteoarthritis; arthritis; arthrodesis; arthroplasty; Gait; step count; walking
MeSH Terms: conditions — Osteoarthritis; Arthritis; Ankylosis | interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimens are used in this project
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Subjects undergoing ankle arthrodesis (fusion) for treatment of ankle arthritis
  Interventions: Procedure: Gait analysis
- Group 2: Subjects undergoing ankle arthroplasty (replacement) for treatment of ankle arthritis
  Interventions: Procedure: Gait analysis

INTERVENTIONS:
Procedure: Gait analysis — Subjects will come into motion analysis laboratory at the VA Puget Sound Health Care System. A standard set of body measurements will be taken using calipers, a measuring tape, and a scale (for example height, weight, leg length, foot length, etc). The investigators will then attach small reflective markers to the body using double-sided tape and ask the participants to walk several times as the motion of each marker is recorded by infrared cameras.

SUMMARY:
The purpose of this study is to determine any functional outcome differences in patients who have undergone surgical treatment for ankle osteoarthritis using surveys, step counts, and laboratory gait analysis.

This study is closed to recruitment; follow-up procedures are completed; the study remains open for data analysis. Enrollment was completed by August 2012.

As of July 2016, the study is currently analyzing data.

In April 2017 the study was approved to begin long term follow-up with study participants. Study personnel contact participants via telephone and/or U.S. Mail to tell them about long term follow-up, and to ask whether they are willing to continue study participation. Long term follow-up will be for up to 12 years after the participant's ankle surgery.

DETAILED DESCRIPTION:
Project Objective:

Ankle osteoarthritis is characterized by joint pain, tenderness, limitation of movement, and variable degrees of inflammation. These factors combined and left untreated will severely limit a person's mobility and willingness to participate in activities. Two common surgical procedures chosen to alleviate pain and to increase mobility are ankle arthrodesis (ankle fusion) and arthroplasty (ankle replacement). Success rates for these procedures are variable and the amount of information available regarding long-term follow-up is limited. The extent to which a person is able and willing to move around the world is often an indicator of his/her condition. The proposed study will examine walking activity levels, and any difference in activity, in patients immediately before and after undergoing surgical treatment for ankle arthritis.

Successfully regaining motility is a priority for patients electing to have surgical treatment for ankle arthritis. A difference in activity levels would indicate an important outcome difference between surgical procedures.

Research Plan:

The investigators propose a mobility outcome study with up to 500 ankle osteoarthritis subjects who will undergo corrective surgery.

Methodology:

The investigators propose a mobility outcome study with a total of up to 500 ankle osteoarthritis subjects before and after surgery over the three years of the study. Ankle arthritis subjects will be recruited from patients at the VA Puget Sound Health Care System (Seattle, WA), Harborview Medical Center (Seattle, WA), Orthopedic + Fracture Specialists (Portland, OR), Orthopaedic Associates of Michigan (Grand Rapids, MN), and Twin Cities Orthopedics (Edina, MN) who have been diagnosed with end stage ankle arthrosis, are ambulatory, speak English, are cognitively intact, and between the ages of 18-80. Recruitment, informed consent procedures and the experimental protocol will be approved by the Institutional Review Board (IRB) at each study site.

Since there is no clinical equipoise it would be unethical to randomize treatment at this time. This project is an observational study of the outcomes following two common treatments: Ankle arthrodesis (fusion) and ankle arthroplasty (total ankle joint replacement). The outcomes will be assessed in two domains:

Functional domain: Each subject's functional status will be determined by the Musculoskeletal Function Assessment (MFA) and the SF-36 general health survey. The MFA is a written questionnaire that assesses activity and social limitations caused by musculoskeletal injury. After completing the questionnaires, subjects will be fit with the Stepwatch Activity Monitor (SAM, Cyma, Seattle WA) around their ankle. An investigator will give them verbal instructions about wearing the SAM. This is a small, pager-sized device which counts the number of steps taken by the wearer. The SAM will be worn around the subject's ankle for 14 days, and then the subject will return the monitor and activity log to the VA by visit or by mail. Assessments using the MFA and SF-36 will occur prior to surgical intervention and at 3, 6, 12, 24, and 36 months following the intervention. Long term follow-up using the MFA and SF-36 was approved in April 2017 and will continue until 12 years after the participant's ankle surgery. Assessments using the SAM will occur prior to surgical intervention and at 3, 6, 12, 24 and 36 months following the intervention. These assessments will provide data on functional limitations due to ankle arthritis and on the efficacy of the treatments in restoring functional ambulation.

Biomechanical domain: Instrumented gait analysis will be performed on each subject. Reflective markers will be placed on each subject's head, hands, arms, trunk, legs, and feet. The subject will walk along a 12 m walkway with embedded forceplates. The motion of the markers will be collected with a 10 camera Vicon 612 system and processed to determine the motion of the ankle joint in three planes as well as the moment and power generated by the ankle during walking. This will allow us to assess the technical functional of the ankle joint, the range of motion used during gait and the moment, power and energy contribution of the ankle during walking for each of the treatments. Gait assessments will occur prior to surgical intervention and at 12, 24, and 36 months post-op. Gait assessment takes place at the VA Puget Sound Health Care System in Seattle, WA. The investigators will only recruit subjects from the VA and Harborview Medical Center for the gait analysis portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Ankle arthritis subjects will be recruited from patients at

  * VA Puget Sound Health Care System (Seattle, WA)
  * Harborview Medical Center (Seattle, WA)
  * Orthopaedic Associates of Michigan (Grand Rapids, MI)
  * Orthopedic + Fracture Specialists (Portland, OR)
  * Twin Cities Orthopedics (Edina, MN)
* who have been diagnosed with end stage ankle arthrosis
* are ambulatory
* speak English
* are cognitively intact
* between the ages of 18-89
* and have elected to undergo surgical correction (arthrodesis or arthroplasty) for end-stage ankle arthritis

Exclusion Criteria:

* Suffer from Rheumatoid Arthritis or other systemic arthritis
* Have any other diseased lower extremity joints or traumatic lower extremity injury that grossly inhibits normal gait

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with ankle osteoarthritis who will undergo either ankle arthrodesis (fusion) or ankle arthroplasty (replacement)
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2025-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J. Sangeorzan, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Segal AD, Cyr KM, Stender CJ, Whittaker EC, Hahn ME, Orendurff MS, Ledoux WR, Sangeorzan BJ. A three-year prospective comparative gait study between patients with ankle arthrodesis and arthroplasty. Clin Biomech (Bristol). 2018 May;54:42-53. doi: 10.1016/j.clinbiomech.2018.02.018. Epub 2018 Mar 5. PMID 29550642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 474 patients were assessed for eligibility with 368 consenting to participate in the study.
  95 subjects were excluded for various reasons (no surgery, non-compliant, etc.) resulting in 273 subjects actively participating.
  229 subjects successively completed the Year 3 follow-up assessment.
Groups:
- Ankle Arthrodesis (Fusion): Subjects undergoing ankle arthrodesis (fusion) for treatment of ankle arthritis
  Gait analysis: Subjects will come into motion analysis laboratory at the VA Puget Sound Health Care System. A standard set of body measurements will be taken using calipers, a measuring tape, and a scale (for example height, weight, leg length, foot length, etc). The investigators will then attach small reflective markers to the body using double-sided tape and ask the participants to walk several times as the motion of each marker is recorded by infrared cameras.
- Ankle Arthroplasty (Replacement): Subjects undergoing ankle arthroplasty (replacement) for treatment of ankle arthritis
  Gait analysis: Subjects will come into motion analysis laboratory at the VA Puget Sound Health Care System. A standard set of body measurements will be taken using calipers, a measuring tape, and a scale (for example height, weight, leg length, foot length, etc). The investigators will then attach small reflective markers to the body using double-sided tape and ask the participants to walk several times as the motion of each marker is recorded by infrared cameras.
Period: Overall Study
Arm/Group | Ankle Arthrodesis (Fusion) | Ankle Arthroplasty (Replacement)
Started | 103 | 170
Completed | 78 | 151
Not Completed | 25 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ankle Arthrodesis (Fusion) | Ankle Arthroplasty (Replacement) | Total
Number analyzed (Participants) | 103 | 170 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (11.4) | 64.4 (9.3) | 61.76 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 81 | 123
  Male | 61 | 89 | 150
Region of Enrollment [Number; unit: participants]
  United States | 103 | 170 | 273

OUTCOME MEASURES:

1. Primary Outcome: Musculoskeletal Functional Assessment (MFA)
Description: Patient reported data using the MFA, a general functional assessment intended as a tool for evaluation of patients' perceptions of their physical, psychological, and social well-being that asks patients to assess their function on 100 items.
  Number shows change in outcome from pre-op to 3 years by surgery type, with a lower score implying an improved outcome (scale range 0 -100.)
Time Frame: Over the course of 3 years
Population: The study started with 103 subjects in the arthrodesis group, and 170 in the arthroplasty group. 78 subjects in the arthrodesis group completed the Year 3 assessment, and 151 in the arthroplasty group. Analysis was done on the MFA data collected from 99 arthrodesis subjects, and 165 arthroplasty subjects.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Ankle Arthrodesis (Fusion): Subjects undergoing ankle arthrodesis (fusion) for treatment of ankle arthritis
- Ankle Arthroplasty (Replacement): Subjects undergoing ankle arthroplasty (replacement) for treatment of ankle arthritis
Arm/Group | Ankle Arthrodesis (Fusion) | Ankle Arthroplasty (Replacement)
Number analyzed (Participants) | 99 | 165
units on a scale | -12.5 (1.4) | -15.0 (0.9)

2. Secondary Outcome: Physical Function Section of Short Form-36 (SF-36)
Description: Patient reported physical function data from the SF-36, a thirty-six item survey evolved from the RAND 36.
  Change in outcome from pre-op to 3 years by surgery type, with a higher score implying an improved outcome (scale range 0 - 100.)
Time Frame: Over the course of 3 years.
Population: The study started with 103 subjects in the arthrodesis group, and 170 in the arthroplasty group. 78 subjects in the arthrodesis group completed the Year 3 assessment, and 151 in the arthroplasty group. Analysis was done on the SF-36 physical function data collected from 93 arthrodesis subjects, and 157 arthroplasty subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ankle Arthrodesis (Fusion) | Ankle Arthroplasty (Replacement)
Number analyzed (Participants) | 93 | 157
units on a scale | 25.4 (2.6) | 31.8 (1.7)

3. Secondary Outcome: Bodily Pain Section of Short Form-36 (SF-36)
Description: Patient reported bodily pain data from the SF-36, a thirty-six item survey evolved from the RAND 36.
  Number shows change in outcome from pre-op to 3 years by surgery type, with a higher score implying an improved outcome (scale range 0 - 100.)
Time Frame: Over the course of 3 years.
Population: The study started with 103 subjects in the arthrodesis group, and 170 in the arthroplasty group. 78 subjects in the arthrodesis group completed the Year 3 assessment, and 151 in the arthroplasty group. Analysis was done on the SF-36 bodily pain data collected from 93 arthrodesis subjects, and 157 arthroplasty subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ankle Arthrodesis (Fusion) | Ankle Arthroplasty (Replacement)
Number analyzed (Participants) | 93 | 157
units on a scale | 35.3 (2.9) | 34.8 (2.0)

ADVERSE EVENTS:
Time Frame: Self-reported outcomes only - no AE reporting included in study.
Arm/Group | Ankle Arthrodesis (Fusion) | Ankle Arthroplasty (Replacement)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was not randomized, and no chart review was conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No